CLINICAL TRIAL: NCT06875245
Title: Comparing Efficacy of 8-Week and 12-Week Faricimab Initial Follow-Up Treatment Intervals Following 4 Loading Doses - Prospective Randomised Study
Brief Title: Comparing Efficacy of 8-Week and 12-Week Faricimab Initial Follow-Up Treatment Intervals
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Martin Pencak, Investigator, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAB 8/12 V1.0
Record Dates: First submitted 2023-10-30; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: retina; amd; faricimab; macula
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — faricimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1, 8-Week (Experimental): Patients in the first group will receive 4 injections of faricimab every 4 weeks, with the next visit and injection after 8 weeks (Week 20 Visit), followed by a treat-and-extend regimen with a minimal interval of 8 weeks and a maximal interval of 16 weeks.
  Interventions: Drug: Faricimab Injection
- Group 2, 12-Week (Experimental): Patients in the second group will also receive 4 loading doses with the next visit after an extended 12-week interval (Week 24 Visit). Following treatment, patients in this group will be on the same treat-and-extend regimen as patients in the first group.
  Interventions: Drug: Faricimab Injection

INTERVENTIONS:
Drug: Faricimab Injection — Intravitreal Injection

SUMMARY:
This is a prospective, randomized study that compares 8-week and 12-week follow-up intervals after the 4 monthly injections in the loading phase. Patients with active CNV confirmed on optical coherence tomography (OCT) and OCT angiography (OCTA) will be randomized into two groups and followed for 44 to 56 weeks.

Patients in the first group will receive 4 injections of faricimab every 4 weeks, with the next visit and injection after 8 weeks, followed by a treat-and-extend regimen with a minimal interval of 8 weeks and a maximal interval of 16 weeks.

Patients in the second group will also receive 4 loading doses with the next visit after an extended 12-week interval. Following treatment, patients in this group will be on the same treat-and-extend regimen as patients in the first group. The study will compare best corrected visual acuity (BCVA), central retinal thickness (CRT) on OCT, and the number of injections between both groups.

DETAILED DESCRIPTION:
Wet age-related macular degeneration (wet AMD) is a progressive eye disease that affects the macula, the part of the retina responsible for sharp central vision. The treatment of wet AMD choroidal neovascularization (CNV) with intravitreal antiVEGF drugs is highly effective. In our study, we aim to compare the efficacy of standard (8 weeks) versus extended follow-up dosing interval (12 weeks) following 4 monthly loading injections of the new combined-mechanism medication, faricimab (6 mg intravitreal dose), which targets both VEGF-A and Ang-2 receptors, in the treatment of wet AMD. We will include all types of CNVs in our study, including Type 1 (occult), Type 2 (classic), Type 3 CNV (Retinal Angiomatous Proliferation = RAP) and mixed CNV. This is a prospective, randomised, comparative study comparing the best corrected visual acuity (BCVA) and central retinal thickness (CRT) on optical coherence tomography (OCT) in the 20th, 24th week of the study between both groups. The total number of injections between both groups will be also compared at the final visit, which will take place between the 44th and 56th week of the study based on the dosing interval.

Patients in the first group will receive 4 injections of faricimab every 4 weeks, with the next visit and injection after 8 weeks (Week 20 Visit), followed by a treat-and-extend regimen with a minimal interval of 8 weeks and a maximal interval of 16 weeks.

Patients in the second group will also receive 4 loading doses with the next visit after an extended 12-week interval (Week 24 Visit). Following treatment, patients in this group will be on the same treat-and-extend regimen as patients in the first group. The study will compare best corrected visual acuity (BCVA), central retinal thickness (CRT) on OCT, and the number of injections between both groups.

Visit plan:

Screening visit - 14 to 0 day prior to baseline. Informed consent will be signed prior to any other study procedures. Ocular and medical history will be written down. BCVA of both eyes will be tested on ETDRS charts. Non-contact intraocular pressure (IOP) will be measured. Slit lamp anterior segment examination and fundus biomicroscopy of both eyes will be performed in artificial mydriasis. The OCT scan of both eyes will be performed, and OCTA will be performed in the treatment naïve eyes. Based on the examination results, patients' eligibility for the study will be assessed.

Baseline - day 1 - BCVA of both eyes will be tested on ETDRS charts. Non-contact IOP will be measured. Slit lamp anterior segment examination and fundus biomicroscopy of both eyes will be performed with artificial mydriasis. OCT of both eyes will be performed. Based on the examination results, patients' eligibility for the study will be assessed. Eligible patients will be randomised, and study medication will be given.

Week 4, Week 8, and Week 12 - adverse events connected to study drugs or study procedures will be assessed and study medication will be given.

Extension Visit Week 20 (group 1) or Week 24 (group 2) - After an initial loading phase of four monthly doses, the two groups differ in the length of the extended dosing intervals. Adverse events connected to study drugs or study procedures will be assessed. BCVA of both eyes will be tested on ETDRS charts. Slit lamp anterior segment examination and fundus biomicroscopy of both eyes will be performed in artificial mydriasis. OCT of both eyes will be performed. Study medication will be given.

Next treatment visit will be scheduled based on the disease activity on the OCT, the ocular examination findings and the BCVA in treat-and-extend regimen with minimal interval of 8 weeks and maximal interval of 16 weeks. The therapeutic interval in both groups may be extended or shortened in up to 4-week increments based on the patient's visual acuity and disease activity, as assessed by OCT evaluating the presence or absence of subretinal or intraretinal fluid or pigment epithelial detachment (PED) and on the presence of other signs of disease activity on the fundus examination (haemorrhage, hard exudates, etc.). It is up to the investigator to make the final decision on the treatment interval.

Follow-up Visits Week 20 to Week 56 - Treat-and-extend regimen. Adverse events connected to study drugs or study procedures will be assessed. BCVA of both eyes will be tested on ETDRS charts. Non-contact IOP will be measured. Slit lamp anterior segment examination and fundus biomicroscopy of both eyes will be performed in artificial mydriasis. OCT of both eyes will be performed. Study medication will be given. Next treatment visit will be scheduled based on the disease activity as described above (treat-and-extend regimen with possible up to 4-week adjustments).

End of Study Visit Week 44-56 - Adverse events assessment. BCVA of both eyes will be tested on ETDRS charts. Slit lamp anterior segment examination and fundus biomicroscopy of both eyes will be performed in artificial mydriasis. OCT of both eyes will be performed. OCTA of the study eye (SE) will be performed.

Study procedures:

OCT - performed on Spectralis OCT (Heidelberg Engineering GmbH, Heidelberg, Germany). CRT will be assessed from automatic retinal thickness analysis in 9 ETDRS subfields including the central subfield. 49 horizontal scans in the angle of 20x20° 123 um apart in High resolution mode with noise reduction set to ART=4 will be performed.

OCTA - performed on Spectralis OCT (Heidelberg Engineering GmbH, Heidelberg, Germany). 512 horizontal scans in the angle of 20x20° 11 um apart in High-speed mode with noise reduction set to ART=5 will be performed.

Disease activity assessment:

Based on the decision of the investigator. Shortening of the treatment interval is recommended when the BCVA decrease of more than 5 ETDRS letters is observed, in case of intra- or subretinal fluid or PED reappearance or increase on the OCT or when new haemorrhage or hard exudates are observed in the macula. Extension of the treatment interval is recommended in the absence of intra- and subretinal fluid and PED on the OCT with better or stable BCVA, or in case the BCVA and OCT findings are stable after 3 injections in the shortest possible interval.

Rescue therapy: Aflibercept may be given as a rescue therapy in case of patients with study drug related sight threatening adverse events or with worsening of BCVA and OCT findings even on the shortest treatment interval when resistance to study drug is suspected. Switch to rescue therapy must be consulted with and approved by principal investigator.

Eligibility

Inclusion criteria:

Active treatment naïve CNV (Type 1, Type 2, or Type 3) in the macula including fovea diagnosed on OCT and OCTA

BCVA between 70 to 35 ETDRS letters (approx. 20/40 to 20/200 Snellen equivalent) decrease in BCVA caused primarily by the CNV in the study eye

presence of intra- or subretinal fluid or PED in the central 1 mm of the macula on the OCT

patient capable of signing the informed consent

Exclusion Criteria:

Myocardial Infarction or Stroke in the last 3 months

Previous or current conditions of the study eye:

1. subretinal haemorrhage comprising more than 25% of the lesion in the study eye
2. scar or fibrosis comprising more than 50% of the lesion in the study eye
3. presence of retinal pigment epithelium (RPE) tears or ruptures in the central 1 mm of the macula in the study eye
4. total lesion size more than 8 papillary diameters (PD) as per OCT and FP examination
5. uncontrolled glaucoma in the study eye defined as IOP of more than 25 mmHg despite the antiglaucoma treatment
6. idiopathic or autoimmune uveitis in the study eye
7. other pathologies in the macula of the study eye unrelated to AMD which can be expected to influence the BCVA (e.g. macular hole, epiretinal membrane, etc.)

k. significant opacities of the ocular media in the study eye including cataract, which can interfere with BCVA assessment or OCT examination

n. diabetic retinopathy, diabetic macular edema or any other retinal vascular disease in the study eye

o. extraocular or periocular infection or inflammation (e.g. blepharitis, keratitis, conjunctivitis, scleritis, etc.) in any eye at the time of screening or baseline visit

p. any intraocular infection or inflammation in any eye during 12 weeks (84 days) before the screening visit

q. allergy or hypersensitivity to any component contained in the study drug

r. pregnant or breastfeeding women

ELIGIBILITY:
Inclusion Criteria:

Active treatment naïve CNV (Type 1, Type 2, or Type 3) in the macula including fovea diagnosed on OCT and OCTA

BCVA between 70 to 35 ETDRS letters (approx. 20/40 to 20/200 Snellen equivalent) decrease in BCVA caused primarily by the CNV in the study eye

presence of intra- or subretinal fluid or PED in the central 1 mm of the macula on the OCT

patient capable of signing the informed consent

Exclusion Criteria:

Myocardial Infarction or Stroke in the last 3 months

Previous or current conditions of the study eye:

1. subretinal haemorrhage comprising more than 25% of the lesion in the study eye
2. scar or fibrosis comprising more than 50% of the lesion in the study eye
3. presence of retinal pigment epithelium (RPE) tears or ruptures in the central 1 mm of the macula in the study eye
4. total lesion size more than 8 papillary diameters (PD) as per OCT and FP examination
5. uncontrolled glaucoma in the study eye defined as IOP of more than 25 mmHg despite the antiglaucoma treatment
6. idiopathic or autoimmune uveitis in the study eye
7. other pathologies in the macula of the study eye unrelated to AMD which can be expected to influence the BCVA (e.g. macular hole, epiretinal membrane, etc.)

k. significant opacities of the ocular media in the study eye including cataract, which can interfere with BCVA assessment or OCT examination

n. diabetic retinopathy, diabetic macular edema or any other retinal vascular disease in the study eye

o. extraocular or periocular infection or inflammation (e.g. blepharitis, keratitis, conjunctivitis, scleritis, etc.) in any eye at the time of screening or baseline visit

p. any intraocular infection or inflammation in any eye during 12 weeks (84 days) before the screening visit

q. allergy or hypersensitivity to any component contained in the study drug

r. pregnant or breastfeeding women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in CRT | from baseline up to 56 weeks
  Change in central subfield thickness (CST) over time as measured by SD-OCT
Patients with intraretinal or subretinal fluid or serous pigment epithelium detachment after loading | From baseline to week 20 (Group 1) or week 24 (Group 2)
  Number of patients with subretinal, intraretinal fluid or pigment epithelium detachment (PED) at week 20 (Group 1) or week 24 (Group 2)

SECONDARY OUTCOMES:
Change from baseline in BCVA | From baseline up to 56 weeks
  Change in best-corrected visual acuity over time as measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters
Presence of fluid | From baseline up to 56 weeks
  Proportion of patients with presence of central retina intraretinal fluid, subretinal fluid, and both at final study visit
Number of injections | From baseline up to 56 weeks
  Number of faricimab injections received during the study duration.
Treatment interval | From baseline up to 56 weeks
  The proportion of patients on a every 4 weeks (Q4w) to every 8 weeks (Q8W), Q8W to every 12 weeks (Q12W), and Q12W to every 16 weeks (Q16W) treatment interval during the study

CONTACTS AND LOCATIONS:
Overall Officials: Martin Pencak, MD, Principal Investigator — +420 267 16 3637
Locations (1):
- Department of Ophthalmology, Faculty hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided